CLINICAL TRIAL: NCT00652860
Title: Chemotherapy, Irradiation, and Surgery for Function-Preserving Curative Therapy of Primary Extremity Soft Tissue Sarcomas: Initial Treatment With I-MAP and GM-CSF; Aerosol GM-CSF During Preoperative Irradiation and Postoperatively
Brief Title: Combination Chemotherapy, Radiation Therapy, and Sargramostim Before and After Surgery in Treating Patients With Soft Tissue Sarcoma That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scott Okuno, M.D., Mayo Clinic
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582297; P30CA015083 (NIH); MC0072 (Other: Mayo Clinic Cancer Center); 1021-01 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-04-03; First posted 2008-04-04 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Metastatic Cancer; Sarcoma
Keywords: lung metastases; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma | interventions — sargramostim; Cisplatin; Doxorubicin; Ifosfamide; Mitomycin; Flow Cytometry; Chemotherapy, Adjuvant; Combined Modality Therapy; Neoadjuvant Therapy; Serotonin Plasma Membrane Transport Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aerosol sargramostim
Biological: sargramostim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: mitomycin C
Other: flow cytometry
Other: immunological diagnostic method
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: multimodality therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: intraoperative radiation therapy
Radiation: selective external radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. GM-CSF may stimulate the immune system in different ways and stop tumor cells from growing. GM-CSF, given by inhalation, may interfere with the growth of tumor cells and prevent metastases from forming. Radiation therapy uses high energy x rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy and GM-CSF before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy and GM-CSF before and after surgery works in treating patients with stage III soft tissue sarcoma that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate 2-year pulmonary metastatic progression rates in patients with primary high-grade extremity soft tissue sarcoma who have received preoperative I-MAP, plus aerosol GM-CSF, plus irradiation with concomitant MAP followed by post-operative aerosol GM-CSF.

Secondary

* To evaluate survival of these patients.
* To evaluate time to progression in these patients.
* To evaluate toxicity in these patients.
* To evaluate tumor response in these patients.

Translational

* To observe and describe sequentially before treatment, after treatment, and after recovery from treatment the frequency of skin test anergy and cellular immunity in extremity soft tissue sarcoma receiving systemic GM-CSF preoperatively and aerosol GM-CSF as part of both preoperative and postoperative treatment.

OUTLINE:

* Neoadjuvant treatment: Patients receive ifosfamide IV over 2 hours on days 0 and 1 and cisplatin IV over 4 hours, mitomycin IV and doxorubicin IV on day 1. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) every 12 hours on days -6 to -3, 2-14, and 22-25. Beginning on day 84 patients also undergo radiotherapy once daily, five days a week, continuing for five weeks. Patients also receive GM-CSF SC twice daily on days -3 and 2 -15 and aerosol GM-CSF twice daily on days 85 - 91, 99 -105, and 113 - 119.
* Chemoradiotherapy: Beginning 4 weeks after completion of neoadjuvant chemotherapy, patients undergo radiotherapy (RT) once daily, 5 days a week, for 5 weeks. Patients also receive aerosolized GM-CSF twice daily on days 2-8, 16-22, and 30-38 and mitomycin C IV, doxorubicin hydrochloride IV, and cisplatin IV over 2 hours on days 1 and 29.
* Surgery: Four weeks after completion of chemotherapy, patients undergo surgery. Patients may also undergo intraoperative RT electron boost or intraoperative high-dose brachytherapy.
* Adjuvant treatment: Beginning 4 weeks after surgery, patients receive aerosol GM-CSF twice daily on days -7, 15-21, 35-42, 56-63, and 77-84. Some patients may undergo external beam RT 2-4 weeks after surgery.

Blood samples are collected at baseline and at 4 and 14 weeks after surgery. Samples are tested for NY-ESO-1 by staining, for T-cell subset by flow cytometry, and for autologous lymphocyte proliferation. Patients may also be tested for delayed-type hypersensitivity and skin test anergy.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and at 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary soft tissue sarcoma

  * Sarcoma must be of the extremity or limb girdle origin
  * No metastatic disease
  * High-grade
* Must be a candidate for preoperative irradiation for potential limb-sparing surgery
* Must not have any of the following:

  * Embryonal rhabdomyosarcoma
  * Extraosseous Ewing sarcomas

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0 - 2
* WBC ≥ 3,500/μL OR granulocyte count ≥1,500/μL
* Platelets ≥150,000/μL
* Direct-reacting bilirubin ≤ 0.3 mg/dL
* Creatinine ≤1.2 times the upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Significant infection
* Active heart disease including any of the following:

  * Myocardial infarction in the past 3 months
  * Symptomatic coronary artery insufficiency
  * First-degree heart block
  * Clinical history of congestive heart failure
* Symptomatic pulmonary disease.

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2001-08; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pulmonary metastatic progression-free rate at 2 years

SECONDARY OUTCOMES:
Survival
Time to progression
Toxicity as per NCI CTC Version 2.0
Tumor response every 4 weeks during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Scott Okuno, MD, Principal Investigator — Mayo Clinic